CLINICAL TRIAL: NCT04726137
Title: European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC) SARS-CoV-2 Antibody Study Protocol
Brief Title: European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC) SARS-CoV-2 Antibody Study Protocol. Covid-19
Acronym: SARS-Cov2
Status: Completed | Type: Observational
Sponsor: PENTA Foundation (Network)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other); University of Athens (Other); University of Cape Town (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Sant Joan de Deu (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Northern Care Alliance NHS Group (Other); University Hospital Birmingham NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); King's College Hospital NHS Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); CHIPS+ Cohort (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17493/002
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Sars-Cov2 Antibodies in Children and Adolescents Living With HIV
Keywords: HIV; COVID-19; Sars-Cov2; children; adolescents; paediatric; cohort; infectious diseases
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scientific knowledge about the COVID-19 pandemic and the virus that is causing it (SARS-CoV-2) is developing rapidly, and the investigators have a clearer idea of the population groups who are at higher risk of becoming infected, having serious illness, and dying. However, less is known about COVID-19 in children, adolescents and young adults living with HIV. It is not yet known whether, or how, HIV affects people's risk of being infected with the virus or becoming ill. This study aims to find out whether children and adolescents living with HIV have had the COVID-19 virus, even if they did not have symptoms and did not realise it at the time.

When a person is infected with a virus, their immune system fights the infection. As a result, they produce proteins called antibodies, and it may take a few weeks for enough antibodies to be made to be detected by a blood test. These antibodies may help protect the person from getting the same infection again. This study wants to find out how many children and adolescents living with HIV across Europe and South Africa have antibodies to the COVID-19 virus. It wants to see if the proportion with antibodies is different in younger children compared to older adolescents and young adults, and whether it varies between different countries.

Children and adolescents with HIV regularly attend hospital outpatient appointments, and during these appointments blood samples may be taken to monitor their health. This study will invite these patients to be tested for antibodies to the COVID-19 virus during their routine visit. The participants will be asked a few short questions about COVID-19 diagnoses in their household and other risk factors for exposure to the virus, and it will collect information on their HIV, medications and any other illnesses they may have. At their next routine clinic visit, approximately 6 months later, it will test them again for antibodies. Testing twice will let see how the percentage of children, adolescents and young adults with antibodies to the COVID-19 virus has changed over time. In South Africa, HIV-uninfected adolescents from a similar socioeconomic background to those living with HIV and recruited to the study will be invited to join this study, which will allow us to compare the prevalence of antibodies across the two groups.

The information from this study will help scientists and healthcare workers care for children, adolescents and young adults living with HIV during the ongoing COVID-19 epidemic in the best possible way. Participants may be given their test results, together with information about what the result means, depending on the usual practice within their clinic.

DETAILED DESCRIPTION:
The study will be conducted within existing cohorts of children, adolescents and young adults living with HIV being followed up in several European countries and South Africa: the European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC) Paediatric Study and the Cape Town Adolescent Antiretroviral Cohort (CTAAC). In CTAAC, adolescents without HIV are also enrolled and will be included in this study. For all participants, two blood samples will be taken at routine clinic visits approximately six months apart and tested for antibodies to SARS-CoV-2; clinical data and data on potential COVID-19 exposures will also be collected.

MAIN AIM OF THE STUDY The overall aim of this study is to describe the prevalence and distribution of antibodies to SARS-CoV-2 in children and adolescents living with HIV in Europe and South Africa.

Primary objective:

•To estimate prevalence of SARS-CoV-2 antibodies in the paediatric and adolescent HIV population and how this changes over time, overall and by key age groups and regions

Secondary objectives:

* To assess factors associated with presence of SARS-CoV-2 antibodies (including demographic factors, antiretroviral treatment, HIV-associated factors or co-morbidities and exposure to household members with COVID-19)
* To estimate the incidence of changes in antibody status to SARS-CoV-2 and associated factors

ENROLMENT Where feasible, all children and adolescents meeting the inclusion criteria and attending the participating clinics during the study period will be invited to take part; where this is not possible, a convenience sample of children and adolescents (e.g. those attending clinic on a specified day of the week) should be invited. The invitation to participate should be independent of the patient's probability of having been exposed to COVID-19. Participants enrolled in the EPPICC Paediatric Study or CTAAC will continue to be followed up as part of the ongoing study.

DATA COLLECTION The study will use data collected in the main EPPICC Paediatric study for participants attending clinics which participate in that study. This includes demographic data and clinical, therapeutic, laboratory and outcome information relating to HIV, COVID-19 and multi-system inflammatory syndrome in children (MIS-C). These data are extracted from clinic records and submitted as part of the main EPPICC study, and will be linked to data collected through the serology study.

Sites which are not members of the EPPICC network will submit equivalent data relating to the time of the two study visits for CLWHIV and HIV-uninfected adolescents.

Additionally, a short questionnaire will be completed by the participant (or their parent / carer) about potential exposures to COVID-19, including diagnoses in household members and known contacts.

For any participant with a record of a suspected or confirmed COVID-19 or MIS-C diagnosis, the cohort will be asked to complete an additional case record form providing details of the diagnosis (e.g. clinical features, hospital admissions, treatments and outcomes).

Cohorts will send pseudonymised electronic datasets to the MRC CTU at UCL. Transfer of data to the MRC CTU at UCL takes place using Galaxkey or an equivalent secure method such as UCL's REDCap server. Data will then be uploaded into a customised database.

LABORATORY TESTING Where sites are conducting serological testing as part of standard care, venous blood samples taken at each site will be transported to the laboratory(ies) routinely carrying out antibody testing for that site. Samples will be analysed with the tests used by each site in routine practice according to manufacturers' instructions or, if in-house tests are used, local SOPs/protocols.

At sites not offering routine serological testing, arrangements should be made with local laboratories for testing. There is strong preference for tests for IgG against the viral spike protein; however, it is recognised that there may be local considerations influencing the range of tests available across settings and results from other tests will be considered.

DISCONTINUATION OR EARLY WITHDRAWAL OF PARTICIPANTS Participants (or their parents/carers) may withdraw from the study at any time without providing a reason.

Participants wishing to withdraw from the study will be offered two options:

1. Participants may withdraw from active follow-up (i.e. future study procedures) within this study but allow the retention and use of data already collected, and further linkage with other data sources as described in the Participant Information Sheet.
2. Participants may withdraw completely from the study, in which case all data and samples collected (if not already tested) would be destroyed and no further follow-up or linkage would take place as part of this study.

Should a participant (or their parent / carer) lose the capacity to consent, they will be withdrawn from active follow-up and their data / samples retained and included in data linkages. Participants who withdraw for any reason will not be replaced.

All withdrawals will be recorded in the study database.

ANALYSIS PLAN Proportions with SARS-CoV-2 antibody at baseline and follow-up and the number/incidence of changes in antibody status between baseline and subsequent test will be estimated overall and by key patient characteristics, region, history of symptomatic COVID-19, contact with COVID-19 cases. Factors associated with the presence of SARS-CoV-2 antibody, changes in antibody status and any subsequent COVID-19 diagnosis (if numbers allow), will be explored using univariable and multivariable logistic and Poisson regression. Exposures of interest include age, sex, ART class and regimen (e.g. protease inhibitor- or tenofovir-based versus other), CD4 count, viral load, ethnicity, BMI-for-age z-score, co-infections (e.g. tuberculosis), co-morbidities and household size.

The association between HIV status and SARS-CoV-2 seropositivity, changes in antibody status and subsequent COVID-19 diagnosis will be assessed in the South African cohort (which includes HIV-uninfected children as well as CLWHIV) using similar methods.

If there is substantial variation in the type of antibody test used (anti-S versus anti-N), analyses will be stratified by type of test. For participants with positive results at both baseline and follow-up and if data allow, quantitative antibody results will be explored to qualitatively describe the possible contribution of re-exposure boosting antibody responses (versus persistence of an existing response).

In sensitivity analyses, we will investigate the implications of misclassification of results due to imperfect sensitivity / specificity of the serological tests used.

COMPLIANCE The study will be conducted in compliance with the approved protocol, the Declaration of Helsinki 1996, the principles of Good Clinical Practice as laid down by the ICH topic E6 (R2), General Data Protection Regulation and the UK Data Protection Act 2018 (DPA number: Z6364106), and the UK Policy Framework for Health and Social Care Research.

Each cohort is responsible for ensuring compliance with local and national regulatory and ethical processes, and data protection.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years at HIV diagnosis
* Current age under 25 years
* Attending routine HIV care in a participating clinic
* Currently in follow-up in CTAAC, a cohort which contributes to EPPICC, or another collaborating cohort
* If aged ≥16 years (or local legal adult age), willing and able to give informed consent to participate in the study
* If aged <16 years (or local legal adult age), a parent/carer able to give informed consent for participating in the study (and, depending on local requirements, those aged ≥10 years, with capacity, to also provide assent).

In addition, in South Africa HIV-uninfected adolescents will be eligible to participate in the study during planned study visits if they meet the following inclusion criteria:

* Current age under 25 years
* In follow-up in the CTAAC study
* If aged ≥18 years, willing and able to give informed consent to participate in the study
* If aged <18 years, a parent/carer is able to give informed consent for participating in the study and participant willing and able to provide assent.

Exclusion Criteria:

Children and adolescents are ineligible if they are taking part in a COVID-19 / SARS-CoV-2 vaccine study at enrollment.

However, should a participant who is enrolled in the EPPICC-SARS-CoV-2 study subsequently join a COVID-19 / SARS-CoV-2 vaccine study or receive a COVID-19 / SARS-CoV-2 vaccine, these are not reasons for exclusion from this study. Data will be collected on vaccine receipt and participation in vaccine studies.

Max Age: 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric infectious disease clinics across Europe and ongoing study in South Africa
Sampling Method: Probability Sample
Enrollment: 906 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Intira J Collins, PhD, Study Director — jeannie.collins@ucl.ac.uk
Locations (7):
- Centre Hospitalier Universitaire Saint Pierre, Brussels, Belgium
- "Agia Sophia" Children's Hospital of Athens, First Department of Paediatrics & Immunobiology & Vaccinology, Athens, Greece
- University of Cape Town, Cape Town, South Africa
- Spain (2):
  - Hospital Sant Joan De Déu, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
- CBO Perinatal Prevention of AIDS Initiative (PPAI), Odesa, Ukraine
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort.: This is an observational study in which consenting participants were enrolled from existing cohorts (EPPICC European Pregnancy and Paediatric Infections Cohort Collaboration, CTAAC Cape Town Adolescent Antiretroviral Cohort and CHIPS+ Collaborative HIV Paediatric Study+). EPPICC and CHIPS+ comprise children and adolescents living with HIV (CALWHIV); CTAAC also enrols HIV-negative adolescents. Participants were eligible if they were aged <25 and, amongst CALWHIV, aged <18 at the time of HIV diagnosis. Initially, SARS-CoV-2 vaccination was an exclusion criterion, although this was subsequently removed in anticipation of increasing vaccine availability. Following informed consent / assent, all participants gave up to two blood samples for serological analysis. (This may be considered as a 'single arm' study).
Period: Overall Study
Arm/Group | Study Cohort.
Started | 906 (Total number of participants recruited.)
Completed | 759 (Total number of participants with two serology test results.)
Not Completed | 147

BASELINE CHARACTERISTICS:
Population: 3 participants were excluded from analysis as they had no valid serology test results
Arm/Group | Study Cohort.
Number analyzed (Participants) | 903
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: One participant was missing age data
  years
    number analyzed (Participants) | 902
    (all) | 17.1 [14.7 to 19.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 476
  Male | 427
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 59
  Black | 612
  Other | 64
  Unknown | 168
Region of Enrollment [Number; unit: participants]
  Greece | 21
  Belgium | 19
  Ukraine | 160
  South Africa | 410
  United Kingdom | 202
  Spain | 91
HIV infection [Count of Participants; unit: Participants] | 800

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Positive SARS-CoV-2 Antibody Test.
Time Frame: Throughout follow-up (at baseline for participants with one sample only; median 6 months for those with two samples)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort.
Number analyzed (Participants) | 903
Participants | 563

2. Primary Outcome: Number of Unvaccinated Participants With at Least One Positive SARS-CoV-2 Antibody Test.
Description: Participants who have not received the SARS-CoV-2 vaccine at the time the sample was taken.
Time Frame: Throughout follow-up (at baseline for participants with one sample only; median 6 months for those with two samples)
Measure: Number; unit: participants
Arm/Group | Study Cohort.
Number analyzed (Participants) | 770
participants | 409

ADVERSE EVENTS:
Time Frame: Throughout follow-up (at baseline for participants with one sample only; median 6 months for those with two samples)
Description: No specific medication was under investigation, data on adverse events and serious adverse events were not collected as part of the study. Data on deaths were captured.
  3 participants were excluded from analysis as they had no valid serology test results.
Arm/Group | Study Cohort.
All-Cause Mortality (participants affected / at risk) | 1/903
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04726137/Prot_SAP_000.pdf